CLINICAL TRIAL: NCT02567955
Title: Immunogenicity and Safety of Gardasil-9 and Cervarix When Administered to 9-10-year-old Subjects According to 0-6 Month Schedule
Brief Title: Immunogenicity and Safety of Gardasil-9 and Cervarix
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HPV 2355
Record Dates: First submitted 2015-10-01; First posted 2015-10-05 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: HPV Vaccines Immunogenicity and Safety
Keywords: HPV vaccines, interchangeable use
MeSH Terms: interventions — Papillomavirus Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immunogenicity two doses of Gardasil-9 (Active Comparator): Subjects will receive two doses of Gardasil-9
  Interventions: Biological: Immunogenicity two doses of Gardasil-9
- Immunogenicity Cervarix and Gardasil-9 (Experimental): Subjects will receive a dose Cervarix and a dose Gardasil-9
  Interventions: Biological: Immunogenicity Cervarix and Gardasil-9

INTERVENTIONS:
Biological: Immunogenicity two doses of Gardasil-9 — Subjects will receive two standard doses of Gardasil-9 (0.5 ml)
  Other Names: HPV vaccine
  Arms: Immunogenicity two doses of Gardasil-9
Biological: Immunogenicity Cervarix and Gardasil-9 — Subjects will receive a standard dose of Cervarix (0.5 ml) and a standard dose of Gardasil-9 (0.5 ml)
  Other Names: HPV vaccine
  Arms: Immunogenicity Cervarix and Gardasil-9

SUMMARY:
A ninevalent HPV vaccine (Gardasil-9) has been recently approved for clinical use. No data on immunogenicity and safety of interchangeable use of the ninevalent and the bivalent vaccine (Cervarix) are available. The main objective of this study is to assess the immunogenicity of ninevalent and bivalent HPV vaccines when administered to 9-10-year-old girls and boys according to 0-6 month schedule.

DETAILED DESCRIPTION:
The proportion of subjects with detectable antibodies and antibody geometrical mean titers to 9 HPV genotypes included in the Gardasil-9 vaccine will be assessed 1 and 6 months post-first dose and 1, 18 and 36 months post-second dose of vaccine.

ELIGIBILITY:
Inclusion Criteria:

* 9-10-year-old girls and boys

Exclusion Criteria:

* previously received an HPV vaccine
* immunosuppressed
* known allergy to a vaccine component

Ages: 9 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 376 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Comparison of proportion of subjects with detectable antibodies to 9 HPV genotypes included in the Gardasil-9 vaccine observed in two study arms | 36 months post-second dose of vaccine
  A Luminex Total IgG assay will be used to assess the presence of antibodies and antibody titers to 9 HPV genotypes included in the Gardasil-9 vaccine. Luminex Units will be used for the antibody titers assessment.

SECONDARY OUTCOMES:
Comparison of tolerability profile of Gardasil-9 and Cervarix | During 5 days after each vaccine dose administration.
  Local and general symptoms observed after each vaccine dose will be assessed by using a standardized diary card. Proportion of subjects who reported local and/or general symptoms will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Équipe de recherche en vaccination, Québec, Canada

REFERENCES:
- [Derived] Gilca V, Sauvageau C, Panicker G, De Serres G, Schiller J, Ouakki M, Unger ER. Long intervals between two doses of HPV vaccines and magnitude of the immune response: a post hoc analysis of two clinical trials. Hum Vaccin Immunother. 2019;15(7-8):1980-1985. doi: 10.1080/21645515.2019.1605278. Epub 2019 Jun 3. PMID 31017850
- [Derived] Gilca V, Sauvageau C, Panicker G, De Serres G, Ouakki M, Unger ER. Immunogenicity and safety of a mixed vaccination schedule with one dose of nonavalent and one dose of bivalent HPV vaccine versus two doses of nonavalent vaccine - A randomized clinical trial. Vaccine. 2018 Nov 12;36(46):7017-7024. doi: 10.1016/j.vaccine.2018.09.057. Epub 2018 Oct 9. PMID 30314913